CLINICAL TRIAL: NCT04144647
Title: The Relationship Between Dual-task Gait Performance, Physical Activity Levels, Sleep and Aging in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LRS-18/19-8994
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-01

CONDITIONS: Healthy; Adults
Keywords: dual-tasking; CANTAB; Gait; Cognition; Sleep; activity
MeSH Terms: conditions — Motor Activity | interventions — Watchful Waiting

STUDY DESIGN:
Intervention Model Description: 100 healthy participants aged between 18-80 years old are recruited for this study.
  All individuals that express interest in this study, will be provided with a Participant Information Sheet (PIS) either by email or hard copy by post.
  All prospective subjects will be screened for matching of inclusion criteria. After a potential participant contacts the PhD student, Ms Viktoria Azoidou, regarding his/her interest in participating in the study, the person will be asked to complete the screening questionnaire via telephone or email as per each individual's preference regarding eligibility criteria. If after screening, a potential participant meets the eligibility criteria, an appointment will be arranged to discuss any concerns or answer any questions participants may have regarding the PIS, then sign the written consent form and be assessed attend the research laboratory for the single testing session.
Masking Description: This is a simple case-controlled study of physiotherapy assessments. It doe snot include masking procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults 18-80 years old (Experimental): Healthy adults 18-80 years old
  Interventions: Other: Single testing session

INTERVENTIONS:
Other: Single testing session — All participants that meet the inclusion criteria, will have to attend the research laboratory at Centre for Human and Applied Physiological Sciences, Shepherd's House, Guy's Campus, King's College London, SE1 1UL to be assessed in a single testing session.
  The testing session will require them to complete some questionnaires regarding balance confidence, psychological state, sleep and physical function and to undertake some simple tests of cognitive function. They will also undertake a brief dynamic balance assessment and the dual-task gait test. The dual-task component involves two cognitive tasks (a numeracy and a literacy task) or auditory task. The gait test will be performed separately and then together with each of two cognitive tasks or auditory task.
  On the day, after the testing, each participant will, also, be provided a physical activity monitor (accelerometer-AX3) to wear on their wrist for 24 hours a day, seven days a week without taking it off.
  Other Names: Observational

SUMMARY:
The co-ordination and control of body segments are integral in providing and maintaining postural stability. It is widely accepted that attentional demands for postural control are placed upon the individual, but these vary according to the nature of the task, the age of the individual and their postural stability. It is thought that divided attention (a technique whereby two tasks are performed at the same time whilst rapidly switching attention between the two tasks) is commonly used when multi-tasking. Divided attention may have important clinical implications to falls risk, in that older adults that experience falls have increased difficulty in switching attention between tasks such as walking and talking. Dual tasking paradigms which present postural and cognitive tasks are often used to test attentional demands for posture control and interference between the two tasks. At present it is not known what impact balance confidence, sleep, activity levels or cognitive ability impact on a person's ability to multi-task when performing complex walking tasks that reflect the complexity of mobilising in real-life situations.

DETAILED DESCRIPTION:
The co-ordination and control of body segments are integral in providing and maintaining postural stability. It is widely accepted that attentional demands for postural control are placed upon the individual, but these vary according to the nature of the task, the age of the individual and their postural stability. It is thought that divided attention (a technique whereby two tasks are performed at the same time whilst rapidly switching attention between the two tasks) is commonly used when multi-tasking. Divided attention may have important clinical implications to falls risk, in that older adults that experience falls have increased difficulty in switching attention between tasks such as walking and talking. Dual tasking paradigms which present postural and cognitive tasks are often used to test attentional demands for posture control and interference between the two tasks. At present it is not known what impact balance confidence, sleep, activity levels or cognitive ability impact on a person's ability to multi-task when performing complex walking tasks that reflect the complexity of mobilising in real-life situations.

The proposed study aims to investigate, in healthy adults aged between 18-80 years old, a) the effect of combining functional gait tasks with different types of dual-tasks and cognitive task categories on total Functional Gait Assessment (FGA) score (primary task), and task prioritisation; b) the relationship between FGA single and dual task performance, age, sleep and PA levels; c) the relationship between age, balance confidence, psychological symptoms and sleep with functional gait single and dual task performance, cognitive function, quality of life and PA levels.

Principle Research Questions:

* What is the effect of dual-task type and/or cognitive task category on FGA performance (primary task), gait speed and task prioritisation?
* What is the relationship between age, balance confidence, psychological symptoms, quality of life and sleep with FGA single and dual task performance, cognitive function and PA levels in healthy adults?

Hypothesis:

1. Cognitive dual tasks will affect performance of the primary FGA task, gait speed and task prioritisation more than an auditory dual task.
2. A more sedentary lifestyle, increasing age, poorer sleep state, balance confidence and/or lower (i.e. poorer performance) cognitive function test scores will affect performance on FGA dual task performance.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling healthy adults
* aged 18-80 years old
* independently mobile.

Exclusion Criteria:

* Individuals have a central nervous system disorder vestibular disorder and/or acute orthopaedic/musculoskeletal disorder affecting balance control and/or gait
* individuals with lack of a good grasp of written and spoken English language.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Functional Gait Assessment | 5 minutes
  The primary outcome is the Functional Gait Assessment which is a 10-item test that assesses performance on complex gait tasks (i.e. walking with head turns, stepping over an obstacle or stopping and turning). Scores range from 0 to 30. The highest score is 30 and greater outcomes are indicative of better performance while lower scores are indicative of poorer performance. The Functional Gait Assessment has been validated in healthy people, older adults with a history of falls and balance impairments, and people with a vestibular disorder. The minimal detectable change for Functional Gait Assessment is reported to be 6 points in persons with balance and vestibular disorders. Scores ≤22/30 identify fall risk and are predictable of falls in community-living older persons within 6 months.

SECONDARY OUTCOMES:
Functional Gait Dual-Task Test | 30 minutes
  The Functional Gait Assessment in isolation will always be completed first in (primary outcome measure), followed by the dual-task test conditions, which will be completed in random order. The cognitive dual-tasking condition will involve a numeracy and literacy task and the auditory stimuli will involve restaurant noise.
Mini-Balance Evaluation Systems Test | 5 minutes
  The Mini-Balance Evaluation Test is a measure of dynamic balance (anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait). The Mini-Balance Evaluation Systems Test consists of 14 items, with scores ranging from 0 to 28 points. Higher scores indicate better outcome while lower scores poorer outcome. Scores ≤ 20/32 indicate increased falls risk.
Cambridge Neuropsychological Test Automated Battery | 45 minutes
  Cambridge Neuropsychological Test Automated Battery is a semiautomated computer program that utilizes a touch screen technology and press pad, to assess neurocognitive function. The Cambridge Neuropsychological Test Automated Battery core cognition battery is a validated cognitive assessment system for assessing multiple components of cognitive function, including attention, visual memory, spatial memory, executive function and reaction time.
Standard pure tone audiometry | 10 minutes
  Standard pure tone audiometry is considered a 'gold' standard test of audiologic examination. This test will be completed with a portable calibrated audiometer (GSI Pello Standard model with DD45's, IP30 and B81, Serial Number: GS0071085, calibrated by Guymark UK Ltd).
Speech in Babble Test | 10 minutes
  The Speech in Babble Test is a low redundancy speech in babble type noise test. The Speech in Babble Test is presented on a calibrated computer using Matlab software. There are 8 in total phonemically and phonetically balanced word lists. The words are presented in the background of a 20-talker babble noise. Two randomly selected monosyllabic consonant vowel consonant word lists in a background of multitalker babble are presented to each ear (i.e. each ear is tested twice). The signal to noise ratio during the test is varied adaptively.
Axivity Wrist Band 3-Axis logging accelerometer | 7 days
  Participants' physical activity level will be assessed using a wrist-worn accelerometer, the Axivity Wrist Band 3-Axis logging accelerometer. The Axivity Wrist Band 3-Axis logging accelerometer captures triaxial acceleration data at 100 Hz with a dynamic range of ±8 g and has been widely used in population-based studies to assess physical activity levels.
Activity-specific Balance Confidence Scale | 3 minutes
  The Activity-specific Balance Confidence Scale is a self-perceived questionnaire with 16 items and assesses balance confidence in daily activities . Scores range from 0 to 100. Higher scores are indicative of better outcome while lower scores indicate poorer outcome. A score ≤67/100 indicate increased falls risk.
Hospital Anxiety and Depression Scale | 3 minutes
  The Hospital Anxiety and Depression Scale, a 14-item scale which assesses non-somatic anxiety and depression symptoms, will also be completed. Scores range from 0 to 21 for each subscale with a score ≥8 proposed for the identification of caseness, for both depression and anxiety. Higher scores are indicative of poorer outcomes.
Pittsburgh Sleep Quality Index | 3 minutes
  The Pittsburgh Sleep Quality Index generates seven component scores: subjective sleep quality, sleep latency, sleep duration habitual sleep efficiency, sleep disturbance, use of sleeping medication, and daytime dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality while lower scores indicate better outcomes. In distinguishing good and poor sleepers, a global Pittsburgh Sleep Quality Index score >5 yields a sensitivity of 89.6% and a specificity of 86.5%.
Epworth Sleepiness Scale | 3 minutes
  The Epworth Sleepiness Scale is a validated and widely used questionnaire exploring daytime sleepiness. It consists of eight questions that are added together to obtain a single number. Higher scores indicate sleeping disorder while lower scores are indicative of better outcomes. Scores range from 0 to 24. The reference range of 'normal' Epworth Sleepiness Scale scores is 0-10 while Epworth Sleepiness Scale scores of 11-24 represent increasing levels of 'excessive daytime sleepiness'.
EQ-5D-5L | 3 minutes
  The EQ-5D-5L is a generic measure of health status for clinical and economic appraisal. The EQ-5D-5L descriptive system comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Situational Vertigo Questionnaire | 3 minutes
  The Situational Vertigo Questionnaire -shortened version measures how frequently symptoms are provoked or exacerbated in environments with visual vestibular mismatch or intense visual motion (e.g. travelling on escalators, crowds, scrolling computer screens). Scores range from 0 to 4. Higher scores indicate poorer outcomes while lower scores are indicative of better outcomes. Scores ≥0.7/4 indicate visual induced dizziness symptoms.
Dizziness Handicap Inventory | 3 minutes
  The Dizziness Handicap Inventory is a 25-item self-assessment inventory designed to evaluate self-perceived handicap imposed by symptoms of dizziness. It consists of three domains: emotional, functional and physical. Total scores range from 0 to 100, with higher score indicating greater perceived handicap while lower scores are indicative of better performance. Scores between 0-30, 31-60, and 61-100 on the Dizziness Handicap Inventory indicate mild, moderate, and severe perceived handicap respectively, and can differentiate a person's functional abilities.
Cognitive and Behavioural Symptom Questionnaire | 3 minutes
  The Cognitive and Behavioural Symptom Questionnaire is a measure of subjects' cognitive (i.e. beliefs) and behavioural responses to symptoms of their health condition. This measure includes five cognitive (i.e. beliefs) subscales: Symptom Focusing, Catastrophizing, Damaging Beliefs, Fear Avoidance and Embarrassment Avoidance; and two behavioural subscales: All or- Nothing and Avoidance/Rest.

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Azoidou, Principal Investigator — King's College London
Locations (1):
- Centre for Human and Applied Physiological Sciences, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participants' data will be processed in accordance with the General Data Protection Regulation 2016 (GDPR). All information collected will be kept strictly confidential and stored anonymously on password protected computers used only by research staff. Data will be stored securely in accordance with the Data Protection Act (1998) and the General Data Protection Regulations which came into effect on 25 May 2018. Participants' data will not be passed on to anyone outside of study research team. Stored, anonymised data may be used for future medical and health-related studies. Data will be retained for 10 years after it has been collected.

REFERENCES:
- [Result] Lacour M, Bernard-Demanze L, Dumitrescu M. Posture control, aging, and attention resources: models and posture-analysis methods. Neurophysiol Clin. 2008 Dec;38(6):411-21. doi: 10.1016/j.neucli.2008.09.005. Epub 2008 Oct 9. PMID 19026961
- [Result] Woollacott M, Shumway-Cook A. Attention and the control of posture and gait: a review of an emerging area of research. Gait Posture. 2002 Aug;16(1):1-14. doi: 10.1016/s0966-6362(01)00156-4. PMID 12127181
- [Result] Yogev-Seligmann G, Hausdorff JM, Giladi N. The role of executive function and attention in gait. Mov Disord. 2008 Feb 15;23(3):329-42; quiz 472. doi: 10.1002/mds.21720. PMID 18058946
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Result] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976
- [Result] Marchetti GF, Lin CC, Alghadir A, Whitney SL. Responsiveness and minimal detectable change of the dynamic gait index and functional gait index in persons with balance and vestibular disorders. J Neurol Phys Ther. 2014 Apr;38(2):119-24. doi: 10.1097/NPT.0000000000000015. PMID 24637931
- [Result] Wrisley DM, Kumar NA. Functional gait assessment: concurrent, discriminative, and predictive validity in community-dwelling older adults. Phys Ther. 2010 May;90(5):761-73. doi: 10.2522/ptj.20090069. Epub 2010 Apr 1. PMID 20360052
- [Result] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Result] Leddy AL, Crowner BE, Earhart GM. Utility of the Mini-BESTest, BESTest, and BESTest sections for balance assessments in individuals with Parkinson disease. J Neurol Phys Ther. 2011 Jun;35(2):90-7. doi: 10.1097/NPT.0b013e31821a620c. PMID 21934364
- [Result] King L, Horak F. On the mini-BESTest: scoring and the reporting of total scores. Phys Ther. 2013 Apr;93(4):571-5. doi: 10.2522/ptj.2013.93.4.571. No abstract available. PMID 23547173
- [Result] Cambridge-Cognition-Limited. CANTABeclipse™: Test Administration Guide Manual. 3rd ed. Cambridge 2015.
- [Result] Egerhazi A, Berecz R, Bartok E, Degrell I. Automated Neuropsychological Test Battery (CANTAB) in mild cognitive impairment and in Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Apr 13;31(3):746-51. doi: 10.1016/j.pnpbp.2007.01.011. Epub 2007 Jan 16. PMID 17289240
- [Result] Fowler KS, Saling MM, Conway EL, Semple JM, Louis WJ. Paired associate performance in the early detection of DAT. J Int Neuropsychol Soc. 2002 Jan;8(1):58-71. PMID 11843075
- [Result] Bamiou DE, Iliadou VV, Zanchetta S, Spyridakou C. What Can We Learn about Auditory Processing from Adult Hearing Questionnaires? J Am Acad Audiol. 2015 Nov-Dec;26(10):824-37. doi: 10.3766/jaaa.15009. PMID 26554488
- [Result] British Society of Audiology. Standard pure tone audiometry. British Society of Audiology-BSA 2017.
- [Result] British Society of Audiology. Standard pure tone audiometry. British Society of Audiology-BSA 2011.
- [Result] Doherty A, Jackson D, Hammerla N, Plotz T, Olivier P, Granat MH, White T, van Hees VT, Trenell MI, Owen CG, Preece SJ, Gillions R, Sheard S, Peakman T, Brage S, Wareham NJ. Large Scale Population Assessment of Physical Activity Using Wrist Worn Accelerometers: The UK Biobank Study. PLoS One. 2017 Feb 1;12(2):e0169649. doi: 10.1371/journal.pone.0169649. eCollection 2017. PMID 28146576
- [Result] Lee IM, Shiroma EJ. Using accelerometers to measure physical activity in large-scale epidemiological studies: issues and challenges. Br J Sports Med. 2014 Feb;48(3):197-201. doi: 10.1136/bjsports-2013-093154. Epub 2013 Dec 2. PMID 24297837
- [Result] Clarke CL, Taylor J, Crighton LJ, Goodbrand JA, McMurdo MET, Witham MD. Validation of the AX3 triaxial accelerometer in older functionally impaired people. Aging Clin Exp Res. 2017 Jun;29(3):451-457. doi: 10.1007/s40520-016-0604-8. Epub 2016 Jul 19. PMID 27435918
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Result] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Result] Guerraz M, Yardley L, Bertholon P, Pollak L, Rudge P, Gresty MA, Bronstein AM. Visual vertigo: symptom assessment, spatial orientation and postural control. Brain. 2001 Aug;124(Pt 8):1646-56. doi: 10.1093/brain/124.8.1646. PMID 11459755
- [Result] Bisdorff A, Von Brevern M, Lempert T, Newman-Toker DE. Classification of vestibular symptoms: towards an international classification of vestibular disorders. J Vestib Res. 2009;19(1-2):1-13. doi: 10.3233/VES-2009-0343. No abstract available. PMID 19893191
- [Result] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Result] Whitney SL, Wrisley DM, Brown KE, Furman JM. Is perception of handicap related to functional performance in persons with vestibular dysfunction? Otol Neurotol. 2004 Mar;25(2):139-43. doi: 10.1097/00129492-200403000-00010. PMID 15021773
- [Result] Skerrett TN, Moss-Morris R. Fatigue and social impairment in multiple sclerosis: the role of patients' cognitive and behavioral responses to their symptoms. J Psychosom Res. 2006 Nov;61(5):587-93. doi: 10.1016/j.jpsychores.2006.04.018. PMID 17084135
- [Result] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Result] Lajoie Y, Gallagher SP. Predicting falls within the elderly community: comparison of postural sway, reaction time, the Berg balance scale and the Activities-specific Balance Confidence (ABC) scale for comparing fallers and non-fallers. Arch Gerontol Geriatr. 2004 Jan-Feb;38(1):11-26. doi: 10.1016/s0167-4943(03)00082-7. PMID 14599700